CLINICAL TRIAL: NCT05451940
Title: Assessing Combination Hydroxyurea and Exogenous Erythropoietin in Sickle Cell Disease
Brief Title: Hydroxyurea and EPO in Sickle Cell Disease
Acronym: ACHiEvE-SCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Julia Xu (Other)
Collaborators: Carnegie Mellon University (Other); American Society of Hematology (Other)
Responsible Party: Sponsor-Investigator, Julia Xu, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120027
Record Dates: First submitted 2022-06-24; First posted 2022-07-11 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anemia, Sickle Cell; Sickle Cell Disease
Keywords: Sickle cell disease; Anemia; Erythropoietin; Hydroxyurea; Sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — Hydroxyurea; Erythropoietin; Hematinics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erythropoietin (Experimental): Subjects on a stable dose of hydroxyurea will be treated with increasing doses of subcutaneous erythropoietin (EPO) as tolerated for an initial 12 weeks, during which the main safety and efficacy endpoints (including the primary endpoint of hemoglobin response) will be assessed. Subjects may continue on treatment for an additional 12 weeks as clinically indicated, with assessment of additional endpoints at the end of the 24-week study period.
  Interventions: Drug: Hydroxyurea; Drug: Epoetin Alfa-BioSimilar

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea is an orally available antimetabolite medication that has been shown to reduce the frequency of painful crises and acute chest syndrome in adults and children with sickle cell disease. Hydroxyurea treats sickle cell disease by a number of different mechanisms, including increasing the expression of fetal hemoglobin (HbF), which reduces sickling of red blood cells.
  Other Names: Droxia, Hydrea, and hydroxycarbamide.
Drug: Epoetin Alfa-BioSimilar — Epoetin alfa and its biosimilars are first-generation erythropoiesis-stimulating agents (ESAs), which are recombinant versions of erythropoietin (EPO) produced using recombinant DNA technology. Erythropoietin (EPO) is a glycoprotein hormone, naturally produced mainly in the kidneys in response to hypoxia and stimulates red blood cell production (erythropoiesis) in the bone marrow.
  Other Names: EPO, epoetin, erythropoietin, erythropoiesis-stimulating agent, ESA, haematopoietin, haemopoietin

SUMMARY:
The proposed study is a Phase 1/2 multi-center study evaluating the safety and efficacy of erythropoietin (EPO) in combination with hydroxyurea in the treatment of chronic anemia in patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a devastating inherited hemoglobin disorder characterized by recurrent episodes of pain and chronic hemolytic anemia. Chronic anemia contributes to multi-organ damage and decreased life expectancy in SCD. However, there are limited treatment options for anemia in SCD. Erythropoietin (EPO) is the standard of care for treatment of anemia related to chronic kidney disease (CKD) and is also used ad hoc in patients with SCD. However, there is limited data on the safety and efficacy of EPO in patients with SCD, especially in combination with hydroxyurea. Therefore, this study aims to treat patients on stable hydroxyurea therapy with subcutaneous EPO, with the goal of assessing the safety of EPO therapy and its effect on chronic anemia in SCD.

(Note: Outcome measure changes were in place prior to study initiation.)

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Confirmed diagnosis of SCD (HbSS or HbS/β0-thalassemia genotypes)
* Screening Hb ≤ 9.0 g/dL
* Screening transferrin saturation ≥ 20% and ferritin ≥ 50 ng/mL
* Must be on stable-dose hydroxyurea treatment (i.e., no changes in dose within 60 days prior to start of study drug) and plan to continue taking hydroxyurea at the same dose and schedule during the study
* If receiving L-glutamine or crizanlizumab, must have been receiving the drug at a stable dose for at least 60 days prior to screening and plan to continue taking the drug at the same dose and schedule during the study

Exclusion Criteria:

* Participating in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes) and/or planning on undergoing an exchange transfusion during the duration of the study; episodic transfusion in response to worsened anemia or VOC is permitted, but participant should not have received a blood transfusion within 60 days of start of study drug
* Received voxelotor or EPO within 30 days of start of study drug
* Untreated iron deficiency, or had initiation or change in dose of supplemental iron within 30 days of start of study drug
* Ongoing acute illness, infection, or VOC within 2 weeks of start of study drug
* Arterial or venous thrombosis within 180 days of start of study drug
* Grade 3 hypertension (defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; medical intervention indicated; more than one drug or more intensive therapy than previously used indicated) on two consecutive measurements
* Unstable angina, uncontrolled seizure disorder, or active malignancy
* End-stage renal disease requiring hemodialysis
* Current pregnancy or breastfeeding
* Received active treatment on another investigational trial within 30 days (or 5 half-lives of that agent, whichever is greater) prior to start of study drug or plans to participate in another investigational drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Z Xu, MD, MScGH, Principal Investigator — University of Pittsburgh
Locations (2):
- UPMC, Pittsburgh, Pennsylvania, United States
- Lagos University Teaching Hospital, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Data collected may be shared with secondary researchers within or outside the participating centers upon request. The shared data will be deidentified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available indefinitely.
Access Criteria: Data use agreement (DUA) may be needed for data to be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will be identified through outpatient hematology clinics at Lagos University Teaching Hospital and UPMC Adult Sickle Cell Clinic. Treating clinicians may refer eligible patients, and study staff may review clinic schedules and electronic health records to identify potentially eligible individuals. IRB-approved recruitment materials may be used, and interested individuals may self-refer by contacting the study team.
Pre-assignment Details: Interested individuals will undergo an informed consent process prior to any study-specific procedures. Eligibility will be confirmed through review of medical history, laboratory values, and other inclusion and exclusion criteria. Participants who meet all eligibility criteria will be enrolled and assigned to the study intervention.
Period: Treatment Period
Arm/Group | Erythropoietin
Started | 17
Completed | 16
Not Completed | 1
Not completed — Physician Decision | 1
Period: Observation Period
Arm/Group | Erythropoietin
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants completing the 12-week treatment period were included in the analysis.
Arm/Group | Erythropoietin
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: Year] — Mean age at enrollment
  Year | 30 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender that participant identifies with at baseline
  Participants
    Female | 9
    Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race that participant identifies with African, Black, or African-American Population: All participants self-identified as African, African-American, or Black
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 16
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-identified as hispanic or non-hispanic
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 16
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Nigeria | 14
  United States | 2
Sickle cell disease genotype [Count of Participants; unit: Participants]
  Hemoglobin SS disease | 16
  Hemoglobin SC disease | 0
  Hemoglobin S/beta0-thalassemia | 0
  Hemoglobin S/beta+-thalassemia | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin (Hb) Response
Description: Hb response is defined as a Hb increase of ≥ 1.0 g/dL at 12 weeks compared to baseline
Time Frame: Baseline to 12 weeks
Population: All enrolled participants who have completed baseline and end of treatment testing, regardless of duration of treatment with EPO, will be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin
Number analyzed (Participants) | 16
Participants | 15

2. Secondary Outcome: Change in Number of Blood Transfusions Per Year
Description: Annualized number of units of simple red blood cell transfusions received in the 12 months before treatment initiation, compared to during the treatment period
Time Frame: Baseline to 12 weeks
Population: All enrolled participants who have completed baseline and end-of-treatment (12-week) testing, regardless of duration of treatment with EPO, will be included in the analysis.
Measure: Mean (Standard Deviation); unit: Transfusions per year
Arm/Group | Erythropoietin
Number analyzed (Participants) | 16
Transfusions per year | -1.1 (3.7)

3. Other Pre Specified Outcome: Changes in Tricuspid Valve Regurgitant Jet Velocity as Assessed by Echocardiography
Description: Changes in tricuspid valve regurgitant jet velocity
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Changes in Cardiac Index as Assessed by Echocardiography
Description: Changes in cardiac index
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Left Ventricular End-diastolic Volume as Assessed by Echocardiography
Description: Changes in left ventricular end-diastolic volume
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Exercise Capacity as Assessed by 6-minute Walk Test With Modified Borg Dyspnea Scale
Description: Changes in 6-minute walk distance and Modified Borg Dyspnea scale (severity of dyspnea during the 6-minute walk test will be measured on a 10-point scale with 0=nothing at all and 10= maximum severity of breathlessness)
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Hemoglobin (Hb)
Description: Mean change in Hb at 12 weeks compared to baseline
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Erythropoietin
Number analyzed (Participants) | 16
g/dL | 3.0 (1.6)

8. Other Pre Specified Outcome: Changes in Absolute Reticulocyte Count
Description: Changes in absolute reticulocyte count
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Lactate Dehydrogenase
Description: Changes in lactate dehydrogenase
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Renal Function
Description: Changes in serum creatinine (and associated eGFR)
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Urine Albumin-to-creatinine Ratio
Description: Changes in urine albumin-to-creatinine ratio
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Total and Indirect Bilirubin
Description: Changes in total and indirect bilirubin
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in Ferritin
Description: Changes in ferritin
Time Frame: Baseline to 12 weeks; Baseline to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study drug initiation to the end of the treatment period (up to 12 weeks)
Arm/Group | Erythropoietin
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin (N=17)
Vaso-occlusive crisis (Congenital, familial and genetic disorders) | 1 (3) — Vaso-occlusive crisis Grade 3 occurred 3 times in one participant. These events were deemed to be unrelated or unlikely related to study intervention because they were within the participant's expected baseline number of vase-occlusive crises.
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Myelodysplastic syndrome Grade 4 was diagnosed by bone marrow biopsy during the study. This participant was being worked up for chronic worsening anemia prior to entering this study, thus, the AE was deemed unrelated to study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin (N=17)
Anorexia (Gastrointestinal disorders) | 1 (1) — Grade 2, unlikely related to study intervention
Cardiac troponin I increased (Cardiac disorders) | 1 (1) — Grade 1, Possibly related
Cholelithiasis (Hepatobiliary disorders) | 1 (1) — Grade 1, unrelated
Conjunctivitis infective (Eye disorders) | 1 (1) — Grade 2, unrelated
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1, unrelated
Dizziness (Nervous system disorders) | 2 (2) — Grade 1, unlikely related; Grade 2, unrelated
Dysgeusia (Nervous system disorders) | 1 (1) — Grade 1, unrelated
Edema limbs (Blood and lymphatic system disorders) | 1 (1) — Grade 1, unrelated
Headache (Nervous system disorders) | 1 (1) — Grade 1, unlikely related
Lung infection (Infections and infestations) | 1 (1) — Grade 3, unrelated
Menorrhagia (Reproductive system and breast disorders) | 1 (1) — Grade 1, unrelated
Neutrophil count decreased (Investigations) | 8 (10) — Grade 1-3, unrelated to study intervention, deemed to be related to hydroxyurea
Pain (General disorders) | 1 (1) — Grade 1, unrelated to study intervention
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — Grade 1 pain in shoulder, unlikely related; Grade 3 pain from leg ulcer, unrelated to study intervention
Palpitations (Cardiac disorders) | 1 (1) — Grade 1, unlikely related to study intervention
Platelet count decreased (Investigations) | 1 (1) — Grade 1, unrelated to study intervention
Priapism (Congenital, familial and genetic disorders) | 3 (3) — Grade 1, unrelated; Grade 2, unrelated; Grade 2, possibly related to study intervention
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1, unrelated to study intervention
Skin infection (Infections and infestations) | 1 (1) — Grade 2, unrelated to study intervention
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3, unrelated to study intervention
Upper respiratory infection (Infections and infestations) | 1 (1) — Grade 2, unrelated to study intervention

LIMITATIONS AND CAVEATS:
The sponsor provided the study drug (EPO) for the duration of the treatment period (12 weeks). However, the sponsor was not able to provide study drug for a longer study, and participants who wanted to continue on EPO treatment during the observation period had to pay out of pocket or get insurance coverage. Thus, most participants had to discontinue EPO after the treatment period. The long-term safety of EPO treatment in patients with sickle cell disease cannot be evaluated from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT05451940/Prot_SAP_000.pdf